## **Cover Page for Statistical Analysis Plan**

| Sponsor-Investigator: | Marshall Holland |
|-----------------------|-------------------------------------|
| NCT Number: | NCT03539081 |
| Unique Protocol ID: | 201605777 |
| Official Title: | Investigating Mechanisms of Human |
| | Spinal Cord Stimulation for Purpose |
| | of Treating Restless Leg Syndrome |
| Date of Document: | 10 May 2023 |

Throughout the study, continuous measures are reported via means and standard deviations. Changes in femoral and brachial artery blood flow during SCS will be examined using two-way repeated measures ANOVA. Missing values for blood flow and MSNA variables will be imputed via marginal sums of squares using a general linear model approach. All analysis will be performed suing SigmaPlot version 13.0 (Systat Software, Inc.), and p-values less than 0.05 will be considered statistically significant for all analyses.